CLINICAL TRIAL: NCT07362446
Title: A Randomised, Double-Blind, Placebo-Controlled, Study of Xolatryp in Patients Presenting With STEMI Undergoing Primary PCI
Brief Title: Prevention of Reperfusion Injury Outcomes Through Effective Cardioprotection Targeting Myocardial Infarction
Acronym: PROTECT-MI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nyrada Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NYR-2A-001
Record Dates: First submitted 2026-01-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction; Reperfusion Injury; AMI; STEMI (ST Elevation MI)
Keywords: STEMI; PCI
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury; ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xolatryp intravenous infusion (Experimental): After randomization, patients receive primary PCI and standard therapy. Patients assigned to the experimental arm also receive Xolatryp, administered as a single, continuous intravenous infusion (i.v.) for 6 hours.
  Interventions: Drug: Xolatryp
- Placebo intravenous infusion (Placebo Comparator): After randomization, patients receive primary PCI and standard therapy. Patients assigned to the placebo arm also recieve a placebo comparator, administered as a single, continuous intravenous (i.v.) infusion for 6 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xolatryp — Patients assigned to the treatment arm recieve Xolatryp administered as a continuous intravenous (i.v) infusion for 6 hours.
  Arms: Xolatryp intravenous infusion
Drug: Placebo — Patients assigned to the placebo comparator arm receive 0.1% of 20% Intralipid in 0.9% normal saline, administered via continuous intravenous (i.v.) infusion for 6 hours.
  Arms: Placebo intravenous infusion

SUMMARY:
This study is open to adults with ST elevation myocardial infarction (heart attack) undergoing primary percutaneous coronary intervention (PCI). The purpose of this study is to determine whether a medicine called Xolatryp is safe and effective in improving cardiac outcomes. One dose of Xolatryp will be tested in this study.

Participants are put into two groups randomly, which means by chance. One group receives a single 6-hour continuous intravenous infusion of Xolatryp and one group receives placebo. Participants are in the study for about 30 days.

Placebo infusion looks like Xolatryp but do not contain any medicine. Participants are followed up via telephone and there is one visit to the study site on day 30.

Heart health is assessed based on the analysis of blood samples, which are collected at the study site, via electrocardiogram (ECG), echocardiogram and cardiac magnetic resonance (CMR) imaging. At the end of the study, the results are compared between the two groups. During the study, the doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Have provided informed consent.
* Male patients aged 40 to 75 years of age.- Female patients aged 55 to 75 years of age, or women aged 40 to 55 years that have no possibility of being pregnant.
* Patient presents with first-time STEMI, scheduled to undergo primary PCI within 6 h of symptom onset and anticipated door to balloon time < 2 h.
* In combination with symptoms consistent with acute MI, patient must demonstrate ST-elevation at the J-point in two contiguous leads.
* Hemodynamically stable including: systolic BP ≥ 90 mmHg, HR 50-120 bpm.
* Killip Class I or II.
* Oxygen saturation ≥ 92% on room air or low-flow oxygen.
* No ongoing VT/VF at enrolment.
* Male participants with female partners of child-bearing potential must be ready and able to use highly effective methods of birth control for at least 7 days following IP administration.

Exclusion Criteria:

* History or ECG evidence of myocardial infarction or cardiomyopathy.
* Prior major cardiac surgery, including but not limited to coronary artery bypass graft surgery (CABG).
* Known contraindication to CMR (e.g. pacemakers, cochlear implants, aneurism clips, claustrophobia, allergy to contrast medium).
* History of clinically significant renal impairment requiring dialysis or an estimated glomerular filtration rate <30 mL/min.
* Estimated or known body weight < 50 kg, > 120 kg at screening.
* Concurrent enrolment in another investigational device or drug trial, or less than 30 days or 5 half-lives of investigational device or drug (whichever is longer), since ending another investigational device or drug trial(s) or receiving other investigational treatment(s). Patients who are participating in non-interventional, purely observational trials can be included.
* Life expectancy of less than 1 year due to non-cardiac pathology in the opinion of the Investigator.
* Any condition or significant clinical abnormality identified at the time of screening that in the judgment of the Investigator or any sub-Investigator would preclude safe completion of the study.
* Known history of hypersensitivity to the investigational drug, or excipients, or do not want to be exposed to soy or egg (including products and derivatives).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | From enrollment up to and including follow-up assessments on Day 30 (end of study)
  Incidence of adverse events (AE) and serious adverse events (SAE) overall. Incidence of AEs and SAEs deemed related to Xolatryp. Incidence of AEs and SAEs deemed cardiac related.

SECONDARY OUTCOMES:
Plasma concentration of Xolatryp during the infusion | Blood samples will be taken for pharmacokinetic (PK) assessment at 4 hours after start of infusion. Where feasible, a sample should be taken at 10 minutes into the infusion.
  Blood sample(s) taken at 4 hours post the start of infusion
ST-segment elevation resolution | pre-PCI ECG and first post procedural ECG
  Comparison between treatment groups of ST-segment elevation resolution calculated from pre-PCI ECG and first post procedural ECG
Cardiac Injury Biomarkers | 48 hours post PCI
  Plasma Troponin I levels calculated as area under the curve (AUC) over 48 hours post PCI
Incidence of Arrhythmias | Telemetry to 48 hours
  Comparison of number of arrhythmias of interest recorded on telemetry (48 hours) between patients treated with Xolatryp vs Placebo. Arrhythmias of interest are sustained ventricular tachycardia (VT), non-sustained ventricular tachycardia (NSVT), and high degree- atrioventricular (AV) block.

OTHER OUTCOMES:
Cardiac Infarct Size | Day 5 (+/- 2 days)
  Volumetric quantification comparison between treatment groups of cardiac infarct size parameters: Acute myocardial infarct size indexed to left ventricular mass, and Myocardial Salvage Index (MSI).
Left Ventricular End-diastolic volume | Day 5
  Left Ventricular End-diastolic volume measurement from CMR will be used to assess cardiac function on Day 5 (+/- 2 days)
Patient Reported Outcomes (PRO) Questionnaire | Day 30 (end of study)
  36-Item Short Form Health Survey (SF-36)
Left Ventricular Ejection fraction | Day 2 and Day 30
  Left ventricular ejection fraction measurement from echocardiogram will be used to assess cardiac function prior to discharge and 30 days post primary PCI
Left Ventricular Volume | Day 2 and Day 30
  Left Ventricular Volume measurement from echocardiogram will be used to assess cardiac function prior to discharge and 30 days post primary PCI
Left Ventricular Function | Day 2 and Day 30
  Left Ventricular Function measurement from echocardiogram will be used to assess cardiac function prior to discharge and 30 days post primary PCI
Fractional shortening | Day 5
  Left Ventricular End-diastolic volume measurement from CMR will be used to assess cardiac function on Day 5 (+/- 2 days)